CLINICAL TRIAL: NCT00050284
Title: Predictors of Immunologic and Clinical Progression in Subjects With CD4+ Cell Counts Greater Than 350 Cells/mm3 Who Discontinue Antiretroviral Therapy
Brief Title: Discontinuation of Antiretroviral Therapy in Patients With Asymptomatic HIV Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5170
Record Dates: First submitted 2002-12-03; First posted 2002-12-04 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Disease Progression; Anti-HIV Agents; Treatment Interruption
MeSH Terms: conditions — HIV Infections; Disease Progression

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether patients who have asymptomatic HIV infection can discontinue antiretroviral therapy (ART) without adverse clinical, virologic, or immunologic consequences. This study will also assess the virologic, immunologic, and clinical outcomes in any patients who restart ART.

DETAILED DESCRIPTION:
Patients who can discontinue ART without a significant loss of virologic or immunologic control and without an increase in clinical events may be spared the expense and adverse effects of treatment. However, the consequences of treatment discontinuation in patients with asymptomatic HIV infections are not well understood. This study will follow the clinical and immunologic progression of HIV infection in patients who have low HIV viral load and preserved CD4+ cell counts at the time ART is stopped.

Patients will fast for at least 8 hours prior to the first study visit. At this visit, blood will be drawn and body measurements will be taken. Patients will then discontinue their ART. Patients taking nonnucleoside reverse transcriptase inhibitors (NNRTIs) will stop taking NNRTIs 48 hours before withdrawing their other ART drugs. Study visits will occur every 4 to 8 weeks for the first year, then every 12 weeks for the second year. Blood will be taken at most visits, and patients will be asked to fast for at least 8 hours prior to Week 12 and 24 visits and again every 6 months. Patients who reinitiate ART for any reason will be registered to Step 2 and followed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* ART with 2 or more drugs for 6 or more months
* CD4+ cell count(s) > 350 cells/mm3 immediately prior to initiation of first ART
* CD4+ cell count > 350 cells/mm3 within 45 days prior to study entry
* Plasma viral load < 55,000 copies/ml within 45 days prior to study entry
* Willingness to discontinue ART at study entry
* Negative serum or urine pregnancy test within 14 days prior to study entry

Exclusion Criteria:

* Pregnancy or breast-feeding
* Systemic cancer chemotherapy, systemic investigational agents, or immunomodulators within 30 days prior to study entry
* Drug or alcohol use or dependence that would interfere with adherence to study requirements
* Illness requiring systemic treatment and/or hospitalization until the patient either completes therapy or has been clinically stable on therapy for at least 30 days prior to study entry
* Chronic medical condition that would have a negative impact on the participation of the patient or would be expected to result in significant use of the medical care system
* History of an HIV-related illness or complication in CDC categories B and C
* Nonadherence to ART
* Active infection with hepatitis B and currently taking adefovir at doses > 10 mg or 3TC and/or TDF

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Skiest, M. D., Study Chair — University of Texas Southwestern Medical Center
Locations (34):
- United States (34):
  - Univ of Southern California, Los Angeles, California
  - Univ of California, San Diego Antiviral Research Ctr, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo County AIDS Program, Stanford, California
  - Santa Clara Valley Med Ctr, Stanford, California
  - Stanford Univ, Stanford, California
  - Willow Clinic, Stanford, California
  - Harbor General/UCLA, Torrance, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ, Chicago, Illinois
  - Cook County Hosp Core Ctr, Chicago, Illinois
  - Rush-Presbyterian / St.Lukes (Chicago), Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - St. Louis Connect Care, St Louis, Missouri
  - Washington Univ (St. Louis), St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - NYU/Bellevue, New York, New York
  - Chelsea Clinic, New York, New York
  - The Cornell Clinical Trials Unit, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Presbyterian Med Ctr- Univ of PA, Norristown, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hosp, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Comprehensive Care Clinic, Nashville, Tennessee
  - Univ of Texas, Southwestern Medical Ctr, Dallas, Texas

REFERENCES:
- [Background] Le Moing V, Chene G, Leport C, Lewden C, Duran S, Garre M, Masquelier B, Dupon M, Raffi F; Antiproteases Cohorte (APROCO) Study Group. Impact of discontinuation of initial protease inhibitor therapy on further virological response in a cohort of human immunodeficiency virus-infected patients. Clin Infect Dis. 2002 Jan 15;34(2):239-47. doi: 10.1086/324354. Epub 2001 Dec 4. PMID 11740714
- [Background] Mocroft A, Youle M, Moore A, Sabin CA, Madge S, Lepri AC, Tyrer M, Chaloner C, Wilson D, Loveday C, Johnson MA, Phillips AN. Reasons for modification and discontinuation of antiretrovirals: results from a single treatment centre. AIDS. 2001 Jan 26;15(2):185-94. doi: 10.1097/00002030-200101260-00007. PMID 11216926
- [Background] Deeks SG, Wrin T, Liegler T, Hoh R, Hayden M, Barbour JD, Hellmann NS, Petropoulos CJ, McCune JM, Hellerstein MK, Grant RM. Virologic and immunologic consequences of discontinuing combination antiretroviral-drug therapy in HIV-infected patients with detectable viremia. N Engl J Med. 2001 Feb 15;344(7):472-80. doi: 10.1056/NEJM200102153440702. PMID 11172188
- [Background] Daar ES, Bai J, Hausner MA, Majchrowicz M, Tamaddon M, Giorgi JV. Acute HIV syndrome after discontinuation of antiretroviral therapy in a patient treated before seroconversion. Ann Intern Med. 1998 May 15;128(10):827-9. doi: 10.7326/0003-4819-128-10-199805150-00005. No abstract available. PMID 9599194
- [Result] Robertson KR, Su Z, Margolis DM, Krambrink A, Havlir DV, Evans S, Skiest DJ; A5170 Study Team. Neurocognitive effects of treatment interruption in stable HIV-positive patients in an observational cohort. Neurology. 2010 Apr 20;74(16):1260-6. doi: 10.1212/WNL.0b013e3181d9ed09. Epub 2010 Mar 17. PMID 20237308